CLINICAL TRIAL: NCT07274501
Title: The Evaluation of the Effect of Music That the Individuals With Moderate Dental Anxiety Have Started Listening to on Their Anxiety Levels While Waiting for Restorative Dental Treatments in the Patient Waiting Room
Brief Title: The Effect of Music That the Individuals With Moderate Dental Anxiety Have Started Listening to While Waiting
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Kıvanc Dulger, Asst Prof, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/24
Record Dates: First submitted 2025-11-15; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Dental Anxiety
Keywords: Dental anxiety; Music; Oxytocin; Cortisol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): In the control group there will be no music listening
- Experimental 1 (Experimental): The music will be listened to only in the waiting room
  Interventions: Behavioral: Music listening in the waiting room
- Experimental 2 (Experimental): The music will be listened to in the waiting room and it will continue during dental treatment
  Interventions: Behavioral: Music listening in the waiting room

INTERVENTIONS:
Behavioral: Music listening in the waiting room — The patients will start to listen to music in the waiting room
  Arms: Experimental 1; Experimental 2

SUMMARY:
It is aimed to evaluate the effect of music listened to in the waiting room on patients with moderate dental anxiety during the restoration of posterior occlusal dental caries on vital signs, cortisol and oxytocin levels of the participants.

DETAILED DESCRIPTION:
The study will be conducted on 90 patients.

30 patients will be in the control group (the group that listens to no music at all), 30 patients will be in the first experimental group (the group that begins listening to music before treatment and will not listen to music during dental treatment), and 30 patients will be in the second experimental group (the group that begins listening to music in the waiting room and continues listening to music during dental treatment).

The study groups will consist of individuals with moderate anxiety who are systemically healthy and free of any disease. Class I occlusal restorations will be placed on permanent posterior teeth. The study groups will consist of individuals over the age of 18, with no systemic disease, and who are not taking any medication. The groups will be arranged so that there is no significant difference between the number of men and women. The individuals will have occlusal caries to be restored. There will be no condition that would prevent the placement of a rubber dam on the teeth. Pregnant women will not be included in the study. Patients who wish to participate will be included in the study on a voluntary basis after being informed about the study. The Modified Dental Anxiety Scale (MDAS) will be used to determine our patients' dental anxiety levels. Each question in the five-question test will be scored from 1 to 5, and the scores will be added together to create a dental anxiety score. The moderate dental anxiety range is between 10 and 18 and is the level generally included in dental anxiety studies. Patients with an appropriate score will be given an appointment for treatment. Before coming in for treatment, individuals will be asked not to have engaged in intense physical exercise and not to have consumed alcohol, smoked, or consumed caffeinated beverages such as coffee. Patients who accept these conditions will sign an informed consent form and provide a medical history (anamnesis) before starting treatment. During treatment, after the application of a local anesthetic without a vasoconstrictor, a rubber dam isolation sheet will be placed, and the treatment will begin. All sterilization procedures will be strictly followed during patient treatment.

Group 1 (Control Group - No Music Before or During Treatment) In the control group, where patients will not listen to any music at all, initial measurements will include salivary cortisol and oxytocin levels, pulse, body temperature, systolic and diastolic blood pressure, and oxygen saturation upon arrival. In the waiting room, the patient will rest for 15 minutes without listening to any music, although headphones will still be worn to control for external auditory stimuli. Just before the treatment begins, salivary cortisol and oxytocin levels, pulse, body temperature, systolic and diastolic blood pressure, and oxygen saturation will be measured again. The headphones will remain on the ears, but no music will be played during the treatment.In the middle of the procedure, after the caries is removed and the cavity is opened, pulse, blood pressure, oxygen saturation, and body temperature will be re-measured.At the end of the treatment, salivary cortisol and oxytocin levels, pulse, body temperature, systolic and diastolic blood pressure, and oxygen saturation will be measured once more. The MDAS will also be administered.

Group 2 (Patients Will Listen to Music Before Treatment Only; No Music During Dental Treatment) In this experimental group, when the patients arrive at the clinic, their baseline salivary cortisol and oxytocin levels, pulse, body temperature, systolic and diastolic blood pressure, and oxygen saturation will be measured. To prevent exposure to other external sounds, patients will be given headphones and asked to listen to music of their choice for 15 minutes in the waiting room to help them relax. Patients will only listen to music in the waiting room; the music will be stopped before the procedure begins, and no music will be played during the treatment, although the headphones will remain in place. Immediately after music listening in the waiting room and just before the treatment starts, the salivary cortisol and oxytocin levels, pulse, body temperature, systolic and diastolic blood pressure, and oxygen saturation will be re-measured. In the middle of the treatment, after the caries is removed and the cavity is opened, pulse, blood pressure, oxygen saturation, and body temperature will be measured again. At the end of the treatment, to compare the dental anxiety level from arrival to post-treatment, salivary cortisol and oxytocin levels, pulse, body temperature, systolic and diastolic blood pressure, and oxygen saturation will be measured as final assessments. Additionally, the MDAS (Modified Dental Anxiety Scale) will be administered again.

Group 3 (Patients Will Listen to Music Before and During Treatment) In this experimental group, patients will start listening to music in the waiting room and continue listening throughout the dental treatment session. Upon arrival, baseline measurements of salivary cortisol and oxytocin levels, pulse, body temperature, systolic and diastolic blood pressure, and oxygen saturation will be taken. Patients will be provided with personal headphones and allowed to listen to music of their choice for 15 minutes in the waiting room to ensure relaxation. Before the procedure begins, salivary cortisol and oxytocin levels, pulse, body temperature, systolic and diastolic blood pressure, and oxygen saturation will be measured again. Patients will continue listening to their selected music through headphones throughout the treatment. In the middle of the treatment, after the caries is removed and the cavity is opened, pulse, blood pressure, oxygen saturation, and body temperature will be re-measured. At the end of the treatment, to assess whether anxiety has decreased compared to the initial visit, final measurements of salivary cortisol and oxytocin levels, pulse, body temperature, systolic and diastolic blood pressure, and oxygen saturation will be taken. The MDAS will also be administered.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy volunteers,
* Clinical diagnosis of at least one occlusal dental caries
* Must have moderate dental anxiety

Exclusion Criteria:

* Unhealthy volunteers
* Teeth with dental cavities in the adjacent teeth where the rubber dam would not be placed
* Dental caries closer than 1 mm to the pulp tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Salivary cortisol level and oxytocin levels | During waiting in the waiting room and dental treatment, an average of one hour
  Change of salivary cortisol and oxytocin levels (before-after)

SECONDARY OUTCOMES:
Heart rate | During waiting in the waiting room and dental treatment, an average of one hour
  The number of pulse will be measured and will be written down in beats per minute (bpm).
Systolic and diastolic blood pressure | During waiting in the waiting room and dental treatment, an average of one hour
  The blood pressures will be measured by blood pressure monitor and will be recorded in mmHg
Body temperature | During waiting in the waiting room and dental treatment, an average of one hour
  It will be measured by body thermometer and will be recorded in degree of Celcius.
Oxygen saturation | During waiting in the waiting room and dental treatment, an average of one hour
  It will be measured by pulse oximeter. It will be recorded as percentage (%)

OTHER OUTCOMES:
Modified dental anxiety questionnaire | During waiting in the waiting room and dental treatment, an average of one hour
  Modified dental anxiety questionnaire will be applied to participants after finishing dental treatment. The scores will be between 5-25. The lower scores will show better results.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University Faculty of Dentistry, Trabzon, Turkey (Türkiye)